CLINICAL TRIAL: NCT06235606
Title: Liposomal Bupivacaine With Standard Bupivacaine Versus Dexmedetomidine With Standard Bupivacaine for Supraclavicular Brachial Plexus Block in Distal Radial Fracture Surgery: a Randomized Controlled Trial.
Brief Title: Liposomal Bupivacaine With Standard Bupivacaine Versus Dexmedetomidine With Standard Bupivacaine
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW24-024
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- To receive supraclavicular BPB using liposomal bupivacaine with standard bupivacaine (Active Comparator): 10ml of 0.5% plain bupivacaine and 10ml of 1.33% liposomal bupivacaine will be injected.
  Interventions: Drug: Bupivacaine Liposome 13.3 Milligrams/Milliliter [Exparel]
- To receive supraclavicular BPB using dexmedetomidine with standard bupivacaine (Active Comparator): 19.5ml of 0.5% plain bupivacaine and 0.5ml (50mcg) of dexmedetomidine will be injected.
  Interventions: Drug: Dexmedetomidine 0.5milligram (50micrograms)

INTERVENTIONS:
Drug: Bupivacaine Liposome 13.3 Milligrams/Milliliter [Exparel] — Bupivacaine liposome is a multivesicular formulation of bupivacaine that allows rapid absorption and prolonged release of bupivacaine.
  Arms: To receive supraclavicular BPB using liposomal bupivacaine with standard bupivacaine
Drug: Dexmedetomidine 0.5milligram (50micrograms) — Dexmedetomidine is a full α₂ adrenergic receptor agonist roughly eight times more selective for the α₂ receptor than clonidine.
  Arms: To receive supraclavicular BPB using dexmedetomidine with standard bupivacaine

SUMMARY:
Brachial plexus blocks (BPB) are commonly used to provide regional anaesthesia for patients undergoing distal radial fracture surgery. Distal radial (DR) fracture surgery is a commonly performed orthopaedic surgery and is usually associated with moderate postoperative pain. Poor postoperative pain control can impair rehabilitation, delay recovery and negatively impact outcomes after surgery. Liposomal bupivacaine (EXPAREL) is a multivesicular formulation of bupivacaine that allows rapid absorption and prolonged release of bupivacaine. Liposomal bupivacaine may provide prolonged analgesia for up to 72 hours after single injection and may therefore achieve greater analgesic efficacy compared to non-liposomal long-acting local anaesthetics. The addition of additive drugs such as dexmedetomidine to regional nerve blocks can also extend analgesia and improve postoperative pain. However, the effect of adding liposomal bupivacaine versus adding dexmedetomidine in regional nerve blocks is not known. In this project, the investigators propose to conduct a randomized controlled trial to investigate the effect of adding liposomal bupivacaine versus dexmedetomidine in the supraclavicular BPB for acute postoperative analgesia. The investigators will also assess longer term secondary outcomes including upper limb functional scores, chronic pain, and health related quality of life.

ELIGIBILITY:
Inclusion criteria

* American Society of Anesthesiologist (ASA) status I-III
* Age 18-90 years old
* Scheduled for distal radial fracture fixation (Open reduction and internal fixation with volar approaching locking plate)
* Patients with informed consent to participate in the study

Exclusion criteria

* Revision surgery
* Previous fractures or surgery in the affected distal radius
* Surgery involving more than the affected arm
* Higher energy and high-grade fracture cases - road traffic accident, fall from height, open fractures, combined distal radius and distal ulna fractures, fractures requiring external fixation, fractures with severe articular comminution or severe metaphyseal extension, comminuted fractures requiring more than a single volar approach incision and a single volar locking plate implant
* Cases with painful conditions affecting the upper limb prior to surgery such as cervical spine, shoulder, elbow, other hand and wrist problems
* Cases with baseline (pre-injury) QuickDASH score worse than 10 out of 100
* Respiratory compromise (requires long term oxygen)
* History of seizures
* Pre-existing neurological disorder/deficit
* Chronic opioid user (3 months or more)
* Presence of chronic pain condition (pain duration over 3 months)
* Alcohol or substance abuse
* Psychiatric illness
* Impaired mental state
* Local infection
* Allergy to analgesic drugs: local anaesthetic drugs, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs), opioids
* Impaired renal function (defined as effective glomerular filtration rate <30ml/min/1.73m2
* Impaired liver function (defined as plasma bilirubin over 34μmol/L; international normalized ratio [INR] ≥1.7, alanine aminotransferase [ALT] over 100U/L, aspartate aminotransferase [AST] over 100U/L)
* Coagulopathy (platelet count <100,000/ml and/or INR ≥1.5) or the use of anticoagulants (not including aspirin) that precludes the use of supraclavicular BPB
* Pregnancy
* Patient refusal for regional nerve blocks
* Patient refusal to join the clinical trial
* Patient unable/unwilling to attend post-op rehabilitation programme

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Weighted area under curve (AUC) pain score at rest | 0-48 hours after surgery
  Pain severity would be rated at rest after surgery using numerical rating scale (NRS) with 0 to 10 where 0=no pain and 10=the worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong